CLINICAL TRIAL: NCT04623372
Title: Immediate Suture or Directed Wound Healing? Comparative Study of Their Respective Values Following a Punch Skin Biopsy (CICAT)
Acronym: CICAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHM-2020/S11/02
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Punch Skin Biopsy
Keywords: skin biopsy; suture; wound healing
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Intervention Model Description: two parallel groups, in a non-inferiority setting, without any pairing or stratification
Who Masked: Outcomes Assessor
Masking Description: One month after the inclusion a photograph of the scar will be taken. This picture will be evaluated by a blind independent investigator without the presence of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suture (Experimental)
  Interventions: Procedure: suture
- Directed wound healing (Experimental)
  Interventions: Procedure: directed wound healing

INTERVENTIONS:
Procedure: suture — suture by separated knots using a non-absorbable 4.0 wire and application of a dry dressing after the punch skin-biopsy
  Arms: suture
Procedure: directed wound healing — application of a dry dressing without any prior suture after the skin biopsy.
  Arms: Directed wound healing

SUMMARY:
The skin punch-biopsies are frequently used technical acts in the current medical practice. However, while these skills are actually easy to perform, the subsequent healing procedure remains still poorly harmonized. Indeed, it usually depends on the physicians personal experiences and some preconceived considerations without any reliable scientific background. This study aims to explore the performances of a directed wound healing behaviour in comparison with the suture.

DETAILED DESCRIPTION:
Because of the lack of reliable scientific data about this topic, the usual behaviours concerning the subsequent healing procedure after a punch skin biopsy remains still poorly defined and harmonized, currently based on the physicians personal experiences and some preconceived considerations. The few studies available in the literature are supporting the assumption that the use of a directed wound healing could be as effective as the widely-used procedure of performing a suture while it does not downgrade the quality of care. However, due to their methodological quality and applicability, they have not led to a substantial modification of the common behaviours. Moreover, the development of some new and the improvement of the former resources could have changed the situation. Therefore, this study aims to bring some recent pragmatic data to assist the implementation of recommendations regarding the attitude to adopt for the healing procedure after a skin punch-biopsy.

The protocol will consist in a monocentric, prospective, randomized and controlled, interventional study. It will be carried out with two parallel groups, in a non-inferiority setting. All the included participants will undergo a skin biopsy using a punch of 4 mm diameter. Then they will either get a suture by separated knots using a non-absorbable 4.0 wire and a dry dressing, either get only a dry dressing. All the subjects will receive a phone call at five days after the skin biopsy in order to collect the self-evaluation of the maximal experienced pain during the healing period. They will also have a single follow-up appointment one month after the inclusion and a photograph of the scar will be taken during this medical consultation. This picture will be evaluated by a blind independent investigator without the presence of the patient.

ELIGIBILITY:
Inclusion Criteria:

* adult person (age greater than or equal to 18 years)
* either hospitalized patient in a conventional or in a day care department, either seen at a medical appointment in Le Mans General Hospital
* person on whom the indication of one or several skin biopsy(ies) using a punch of 4 mm diameter has been established
* affiliated or beneficiary of a statutory social insurance scheme
* free and informed written consent, signed by both the participant and the investigator (the day of inclusion at the latest and prior to any examination needed by the protocol) after an oral and written information

Exclusion Criteria:

* skin biopsy on the face or the cervical area
* pregnant, breastfeeding or parturient woman
* person deprived of liberty by an administrative act or a court decision
* patient requiring compulsory mental health care
* minor or legally protected adult
* patient that is no longer in a condition to express his or her wishes
* person that have participated or that are taking part in an interventional study over the past 30 days (condition of exclusivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Assess aesthetic quality of the scar by physician | one month after skin punch biopsy
  the asserted aesthetic quality of the scar will be assessed by a dermatologist with 4-level scale

SECONDARY OUTCOMES:
Assess aesthetic quality of the scar by patient | 1 month after skin biopsy punch
  The asserted aesthetic quality of the scar will be assessed by the participant himself using a 4-level scale
Assess maximal pain experienced by the patient | 1 month after skin biopsy punch
  The maximal pain experienced by the patient during the Healing phase will be assessed with a numerical scale ranging from 0 to 10
Assess amount of bleeding | immediately after skin biopsy punch
  the scoring of the amount of bleeding subsequent to the skin biopsy will be assessed with a numerical scale ranging from 0 to 10
Assess clotting time | immediately after skin biopsy punch
  The clotting time subsequent to the skin biopsy will be assessed using a 4-level scale
Observe cutaneous infection | 1 month after skin biopsy punch
  occurrence of a cutaneous infection that had required an antibiotic treatment and/or the achievement of a drainage during the month following the skin punch-biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France